CLINICAL TRIAL: NCT02339909
Title: Incentives in Diabetic Eye Assessment by Screening (IDEAS) Trial
Brief Title: Incentives in Diabetic Eye Assessment by Screening
Acronym: IDEAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: REC 14/LO/1779
Record Dates: First submitted 2014-12-15; First posted 2015-01-16 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetic Retinopathy
Keywords: Screening; Incentives
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): The intervention for the "Control" group consists of the standard invitation letter from the Screening service. (The trial is testing the impact of the different invitation letters on the primary outcome of screening attendance.)
  Interventions: Behavioral: Control
- Fixed Incentive (Experimental): The intervention for the "fixed incentive" group consists of the standard invitation letter from the Screening service, with additional text offering a fixed financial incentive (£10) if they attend screening. (The trial is testing the impact of the different invitation letters on the primary outcome of screening attendance.)
  Interventions: Behavioral: Fixed financial incentive
- Probabilistic Incentive (Experimental): The intervention for the "probabilistic incentive" group consists of the standard invitation letter from the Screening service, with additional text offering a probabilistic financial incentive (entry into a lottery offering at least a 1 in 100 chance to win £1000) if they attend screening. (The trial is testing the impact of the different invitation letters on the primary outcome of screening attendance.)
  Interventions: Behavioral: Probabilistic financial incentive

INTERVENTIONS:
Behavioral: Fixed financial incentive — Participants receiving the "fixed financial incentive" intervention will be sent a screening appointment letter offering them a fixed amount of £10 if they attend their screening appointment.
  Arms: Fixed Incentive
Behavioral: Probabilistic financial incentive — Participants receiving the "probabilistic financial incentive" intervention will be sent a screening appointment letter offering them an entry into a lottery with at least a 1 in 100 chance of winning £1000 if they attend their screening appointment.
  Other Names: Lottery to financial incentive
  Arms: Probabilistic Incentive
Behavioral: Control — Participants receiving the "active comparator", (i.e. "control") intervention, will be sent the standard diabetic retinopathy screening appointment letter.
  Arms: Control

SUMMARY:
This trial is a randomised controlled trial to assess whether annual attendance rates at diabetic eye screening appointments in Kensington, Chelsea and Westminster could be improved by offering invitees a small financial incentive. The research questions are:

1. Are incentives an effective strategy to encourage participation in the screening programme?
2. Does the design of the financial incentive scheme affect its effectiveness in influencing participation in health screening?
3. Does the choice of incentive scheme, if successful, attract patients who have a different demographic or socioeconomic status to those who attend screening regularly?
4. Is offering these incentives a cost-effective strategy for enhancing participation?

DETAILED DESCRIPTION:
An increasing emphasis is being placed on preventative healthcare in the NHS (National Health Service). Screening programmes currently exist in many clinical areas including diabetic retinopathy as well as breast cancer, cervical cancer and cardiovascular disease. In many contexts the benefits of health screening are well documented, but concerns exist about the effectiveness and cost-effectiveness of such programmes as uptake to screening may be very poor in some, generally hard to reach, communities. There are many ways of trying to encourage participation in health promoting activities and it is likely real shifts in behaviour will only come about with a mix of strategies. In this study we set out to see if we can improve screening rates in London, which has both high and low levels of deprivation and specific populations with poor attendance. The ultimate success of a high-quality screening program depends on the uptake rate of the population and novel solutions are required to meet the challenge of achieving this.

Diabetes is an increasing public health concern worldwide. There are 2.9 million people diagnosed with diabetes in the UK (United Kingdom) and an estimated 850,000 people who have the condition but are not recognised. Whilst the rates of other vascular risk factors such as hypertension, smoking and hypercholesterolaemia are falling, the rates of diabetes in the UK are rising. This is despite the co-ordinated efforts of primary and secondary care prevention programmes.

All patients with diabetes are at risk of developing diabetic retinopathy. This condition is caused by the microscopic damage to small blood vessels to the eye. There is proliferation (growth) of these vessels and these new fragile vessels may bleed and destroy the retina leading to sight loss. It is estimated that in England every year 4,200 people are at risk of blindness caused by diabetic retinopathy and there are 1,280 new cases of blindness caused by diabetic retinopathy. It is the leading cause of sight loss in the UK in the working population and therefore there is a significant social and financial burden associated with the condition. However with timely diagnosis and treatment the risk of blindness can be dramatically reduced. As this condition may well remain silent until catastrophic late manifestations of the disease are evident, the need for an effective screening programme is obvious.

The National Screening programme was implemented in England between 2003 and 2006. This involves an annual retinal digital photographic screening offered to all people aged 12 years and older diagnosed with type 1 and type 2 diabetes. The test involves administration of eye drops to the eye and a photograph of the retina taken without contact with the eye. The success of this screening programme is without contest. In 2011-2012, 2,587,000 people in England aged 12 and over were identified with diabetes and over 90% were offered screening for diabetic retinopathy. 1,911,000 received screening which equates to an uptake of 81%. However there is significant variability in uptake in differing areas.

Although screening is offered in multiple locations including GP (general practice) surgeries and hospitals, the poor uptake of screening in socially deprived areas is well documented. For example, in Gloucestershire, with each increasing quintile of deprivation, diabetes prevalence increases (odds ratio 0.84), the probability of having been screened for diabetic retinopathy decreases (odds ratio 1.11), and the prevalence of sight-threatening diabetic retinopathy among screened patients increases also (odds ratio of 0.98).

Since the effectiveness of any screening programme is intimately linked to the uptake by the population (and in particular uptake by those most at risk), simple, inexpensive and cost effective strategies are required by the NHS to influence population health behaviours in domains where choices are often in sharp contrast to underlying intentions. This has relevance to diabetic retinopathy screening but also more widely as we increasingly try to prevent disease rather than simply treat it.

Incentives are central to economics and are used across the public and private sectors to influence behaviour. Psychological phenomena from behavioural economics allow us to design incentive-based interventions that are more effective at delivering improved outcomes. Personal incentives have been used to motivate patients and general populations to change their behaviour. Examples of behaviours targeted include smoking and drug use cessation. Incentives can include cash, vouchers or benefits-in-kind and they can have a profound effect on individual behaviour at a relatively small cost. Interest in offering incentives to foster healthier lifestyles has increased, as the full economic and social costs of bad choices and unhealthy behaviour have become apparent. Incentives have previously been used to improve cancer screening rates, but they have been targeted at the providers of the service rather than people invited to attend for screening. Financial incentives have been seen to be more effective in increasing performance of infrequent behaviours (e.g. vaccinations) rather than in more sustained behaviours (e.g. smoking). As screening usually requires discrete one-off behaviours, incentives may be particularly effective in increasing their uptake.

A wider use of incentives in public health interventions is a more recent phenomenon and has attracted controversy and concerns about whether they are effective (and cost effective) or not. This study will provide evidence to policy makers about the role of different incentive schemes in encouraging health promoting behaviours. We do not suggest that providing incentives is the only answer to encouraging screening participation, but if we demonstrate good evidence that they are effective (and cost effective), their targeted application may be indicated. Equally demonstration that incentives of this type are not effective may prevent unnecessary financial loss from the NHS if wider rollout of such programmes is considered.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients who were invited to screening in the last 24 months on a yearly basis and failed to attend or contact the screening service to rearrange an appointment

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1051 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Bicknell, Principal Investigator — Imperial College London

REFERENCES:
- [Background] Scanlon PH, Carter SC, Foy C, Husband RF, Abbas J, Bachmann MO. Diabetic retinopathy and socioeconomic deprivation in Gloucestershire. J Med Screen. 2008;15(3):118-21. doi: 10.1258/jms.2008.008013. PMID 18927093
- [Background] Marteau TM, Ashcroft RE, Oliver A. Using financial incentives to achieve healthy behaviour. BMJ. 2009 Apr 9;338:b1415. doi: 10.1136/bmj.b1415. No abstract available. PMID 19359291
- See also: Diabetes UK — https://www.diabetes.org.uk/diabetes-the-basics
- See also: NHS diabetic eye screening website — https://www.nhs.uk/conditions/diabetic-eye-screening/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the nature of the study, informed consent could not be collected. The number of participants Started in the Participant Flow (1274) refers to the number randomised. Following randomisation, but prior to being sent the intervention letter, 223 participants became ineligible, so 1051 participants were actually enrolled in the study.
Period: Overall Study
Arm/Group | Control | Fixed Incentive | Probabilistic Incentive
Started | 524 | 375 | 375
Completed | 435 | 312 | 304
Not Completed | 89 | 63 | 71
Not completed — Became ineligible after randomisation | 89 | 63 | 71

BASELINE CHARACTERISTICS:
Population: The number of patients sent letters.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Fixed Incentive | Probabilistic Incentive | Total
Number analyzed (Participants) | 435 | 312 | 304 | 1051
Age, Customized [Count of Participants; unit: Participants]
  16-65 years | 229 | 173 | 176 | 578
  Over 65 years | 206 | 139 | 128 | 473
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 142 | 128 | 442
  Male | 263 | 170 | 176 | 609
Region of Enrollment [Number; unit: participants]
  United Kingdom | 435 | 312 | 304 | 1051

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Attending Screening Appointment
Description: The participants will be invited to a specific appointment between three months and one year from their previous missed appointment. The primary outcome refers to the number of participants who did attend their appointment.
Time Frame: At designated appointment date (between three months and one year from previous missed appointment)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Fixed Incentive | Probabilistic Incentive
Number analyzed (Participants) | 435 | 312 | 304
Participants | 34 | 17 | 10

2. Secondary Outcome: Number of Patients Requiring Intervention After Sight Outcome From Diabetic Retinopathy Screening.
Description: The outcome measure from screening is an ordinal measure indicating whether there is no retinopathy, or varying degrees of retinopathy. This will be measured at the screening appointment (for those participants who attend their appointment). We report whether there is further management required as a result of screening.
Time Frame: Number of patients with additional management triggered as a result of test at designated screening appointment (between three months and one year)
Population: These are the numbers of each group that attended screening and had retinopathy screening
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Fixed Incentive | Probabilistic Incentive
Number analyzed (Participants) | 34 | 16 | 10
Participants | 6 | 7 | 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | Fixed Incentive | Probabilistic Incentive
Serious Adverse Events (participants affected / at risk) | 0/435 | 0/312 | 0/304
Other Adverse Events (participants affected / at risk) | 0/435 | 1/312 | 0/304
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=435) | Fixed Incentive (N=312) | Probabilistic Incentive (N=304)
Patient invited and not suitable for screening (Investigations) | 0 (0) | 1 (1) | 0 (0) — Patients invited and attending, who are not suitable for screening are considered an adverse event in this trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No